CLINICAL TRIAL: NCT07262008
Title: Sustained Mood Improvement With Laughing Gas Exposure: A Randomized Controlled Double-Blind Trial
Brief Title: Sustained Mood Improvement With Laughing Gas Exposure
Acronym: SMILE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Anesthesia Clinical Trials Unit (Department of Anesthesia and Pain Management) (Unknown); University Health Network, Toronto (Other); Sunnybrook Health Sciences Centre (Other); Unity Health Toronto (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Karim Ladha, MD MSc FRCPC, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5428-CTO
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Nitrous Oxide; Midazolam

STUDY DESIGN:
Intervention Model Description: This study will be a phase III, double-blind, randomized, active placebo-controlled, superiority trial with two parallel arms.
Who Masked: Participant, Outcomes Assessor
Masking Description: As noted above, only the individual administering the intervention will be aware of allocation assignment due to safety. The participant and outcomes assessors will be blinded to minimize bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Nitrous oxide+ intravenous Saline
  Interventions: Drug: Inhalation of Nitrous oxide (Laughing gas) + intravenous saline
- Active Control Group (Active Comparator): 100% oxygen+ intravenous midazolam
  Interventions: Drug: inhalation of %100 oxygen + intravenous midazolam

INTERVENTIONS:
Drug: Inhalation of Nitrous oxide (Laughing gas) + intravenous saline — Nitrous oxide at an inspiratory concentration of 50% with concurrent intravenous saline (20ml) for one hour.
  Other Names: Nitrous oxide
  Arms: Intervention Group
Drug: inhalation of %100 oxygen + intravenous midazolam — Inspiration of 100% oxygen with concurrent intravenous midazolam (0.02mg/kg, up to 2 mg) for one hour.
  Other Names: Midazolam
  Arms: Active Control Group

SUMMARY:
Multi-centre, parallel group, blinded, 1:1 randomized controlled trial to determine the effect of nitrous oxide on reducing symptoms of depression in patients with treatment resistant depression.

DETAILED DESCRIPTION:
SMILE is a multi-centre, parallel-group, blinded randomized controlled trial of 120 patients with treatment resistant depression. Consented eligible patients will be randomized to 1) Inhalation of Nitrous Oxide + Intravenous Saline (intervention Group)or 2) Inhalation of Oxygen + Intravenous Midazolam (Active Control Group). Participants will receive their respective study intervention once a week for four weeks for a total of four sessions. Follow-up visits will be conducted over the phone 2-weeks, 4-weeks, and 12-weeks following the last intervention visit. Questionnaires will be administered to assess change in depressive symptoms, function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years of age
2. Meeting Diagnostic and Statistical Manual for Mental Disorders (DSM-5) criteria for Major Depressive Disorder (MDD)
3. Current major depressive episode as confirmed by the Mini International Neuropsychiatric Interview (MINI) for DSM-5
4. Experiencing moderate to severe depressive episodes, as defined by the Montgomery-Åsberg Depression Rating Scale (MADRS) > 21
5. Failure of two trials of antidepressant therapy of adequate dose and duration, during the current depressive episode
6. For women of childbearing potential, use of highly effective or double-barrier methods of contraception. Abstinence is acceptable if it is the preferred and usual lifestyle of the female participant
7. Capacity to provide informed consent.

Exclusion Criteria:

1. Acute suicidality defined as score > 4 on MADRS item 10
2. Diagnosis of Bipolar Disorder
3. Current substance abuse or dependence and/or history of alcohol abuse or dependence within the past year
4. Dementia
5. Current or lifetime history of schizophrenia or schizoaffective disorder
6. Known history of hypersensitivity or allergy to nitrous oxide, midazolam or any ingredients in the study formulations
7. Contraindication to receiving nitrous oxide (e.g. any condition where air is entrapped within a body and its expansion might be dangerous such as, pneumothorax, elevated intracranial pressure, air embolism, recent middle ear, vitreoretinal or bowel obstruction surgeries, etc.)
8. Known chronic cobalamin or folate deficiency (e.g. signs of anemia or neurological symptoms, with plasma levels of homocysteine over 15 µmol/L and abnormal red blood cells and leukocytes on a complete blood count CBC) or current methotrexate use
9. Contraindication to receiving the placebo midazolam (e.g. shock, chronic heart failure, chronic obstructive pulmonary disease, closed-angle glaucoma, renal failure, patients with limited pulmonary reserve or those with severe decline of vital signs)
10. Daily use of centrally acting medicinal products, such as opioid agonists, (e.g. naloxone and naltrexone) morphine derivatives (e.g. oxycodone, hydrocodone, oxymorphone, codeine), benzodiazepines (e.g. diazepam, clonazepam, alprazolam) and/or other central nervous system depressants such as barbiturates (e.g. phenobarbital, pentobarbital, amobarbital) and alcohol within the past week.
11. Pregnancy or breastfeeding
12. Received electroconvulsive therapy within the past six months
13. Received ketamine treatment within the past six months
14. Received repetitive transcranial magnetic stimulation within the past six months
15. Unwilling to maintain current antidepressant regimen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) score | Baseline to the 2-week follow-up (Visit 6 - Day 35).
  The MADRS is a 10-item clinician-rated scale used to assess the severity of depressive symptoms and to detect changes over time in response to treatment. It is commonly used in randomized controlled trials due to its sensitivity to change and strong psychometric properties. The MADRS is also recognized by regulatory and health technology assessment agencies, including the U.S. Food and Drug Administration (FDA) and the Canadian Agency for Drugs and Technologies in Health (CADTH), as an established measure for evaluating treatment efficacy in depression.
  Higher scores indicate worse outcomes and greater severity of depression.

SECONDARY OUTCOMES:
Proportion of patients who achieved a response | 2-week and 12-week follow-ups post last intervention visit
  Defined as a 50% reduction in MADRS score between baseline and the 2- and 12-week follow-ups.
Proportion of patients who achieved remission | 2-week and 12-week follow-ups post last intervention visit
  Defined as achieving both a response and a MADRS score <10 at the 2- and 12-week follow-ups.
Change in self-reported depressive symptoms | 2-week and 12-week follow-ups post last intervention visit
  Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-SR-16) Higher scores are associated with increased severity in depressive symptoms Total scores range from 0-27
  Normal/No Depression 0-5 Mild Depression 6-10 Moderate Depression 11-15 Severe Depression 16-20 Very Severe Depression 21-27
Change in cognitive function | 2-week and 12-week follow-ups post last intervention visit
  Assessed using the Digit Symbol Substitution Test (DSST) The Digit Symbol Substitution Test (DSST) measures processing speed, attention, and executive function by assessing a person's ability to quickly and accurately pair numbers with symbols according to a key. To score it, the total number of correct symbol-for-number substitutions completed within a timed period (typically 90-120 seconds) is counted.
  Higher scores indicate better performance.
Change in functioning and disability | 2-week and 12-week follow-ups post last intervention visit
  Assessed using the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0)
  Total Score Range: 0-100 0 = No disability 100 = Full disability
  WHODAS 2.0 scores reflect overall functioning across six domains (cognition, mobility, self-care, getting along, life activities, and participation).
  Higher scores indicate greater functional impairment.
Change in anxiety symptoms | 2-week and 12-week follow-ups post last intervention visit
  Assessed using the Generalized Anxiety Disorder 7-item scale (GAD-7) A GAD-7 score is interpreted based on its total score, with the range being 0-21, where higher scores indicate more severe anxiety. The standard interpretation is: 0-4 (minimal anxiety), 5-9 (mild anxiety), 10-14 (moderate anxiety), and 15-21 (severe anxiety)
Change in quality of life | 2-week and 12-week follow-ups post last intervention visit
  Assessed using the EuroQoL 5-Dimension 5-Level scale (EQ-5D-5L) The EQ-5D-5L is a standardized, participant-reported measure of health-related quality of life. It assesses five dimensions-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression-each rated across five levels of severity (no problems to extreme problems). Responses are converted into a single index score, typically ranging from <0 (health states worse than death) to 1.0 (full health).
Assessment of Safety via FIBSER Scale | Baseline to Week 12
  Safety outcomes will be assessed by evaluating adverse events in both general and specific terms using the Frequency, Intensity, and Burden of Side Effects Rating (FIBSER) scale.
  FIBSER ; higher score indicates worse outcomes. Clinical Relevance of Question 3: 0-2 = no changes needed; 3-4 = side effects should be addressed; 5-6 = change treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Ladha, MD, Principal Investigator — Women's College Hospital
Locations (5):
- Canada (5):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital (Unity Health), Toronto, Ontario
  - Toronto General Hospital (UHN), Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Toronto Western Hospital (UHN), Toronto, Ontario

REFERENCES:
- [Background] Ladha KS, Lee J, Mattina GF, Pazmino-Canizares J, Wijeysundera DN, Nezhad FG, Tassone VK, Adamsahib F, Lou W, Kennedy S, Bhat V; SMILE Study Investigators. Sustained mood improvement with laughing gas exposure (SMILE): a randomised, placebo-controlled pilot trial of nitrous oxide for treatment-resistant depression. BJPsych Open. 2025 Sep 12;11(5):e208. doi: 10.1192/bjo.2025.10823. PMID 40936464